CLINICAL TRIAL: NCT04300205
Title: High Intensity LED Photobiomodulation (PBM) Therapy for Chronic Leg and Foot Ulcers
Brief Title: High Intensity LED Photobiomodulation Therapy for Chronic Leg and Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illumacell Inc. (Industry)
Collaborators: Kerber Applied Research (Unknown); Alberta Health Services - Lower Limb Wound Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCAB-89340
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot ulcer; venous foot ulcer; phototherapy; photobiomodulation; LED light
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Participants with chronic foot and leg ulcers less than 8 cm in diameter (longest direction) will randomized into one of 2 groups for this study: 1) to receive a free 10 minute light treatment with the KPTL10 device in addition to standard care, or 2) strictly be a part of the standard care control group (no light treatment). For treatment, the light device is placed at a fixed distance (1 cm) above the wound. All participants will have wound measurements taken with digital software throughout the course of the study to track wound healing. Patients will also record their pain levels by filling out a VAS pain scale throughout the study.
Who Masked: Participant
Masking Description: Participants wear black-out glasses during LED phototherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity LED light treatment (Experimental): Participants treated with high intensity LED phototherapy
  Interventions: Device: High intensity LED light device
- Sham high intensity LED light treatment (Experimental): Participants set up to be treated with light device but after being masked, the device is moved off the wound
  Interventions: Device: Sham LED light device

INTERVENTIONS:
Device: High intensity LED light device — Participant wounds are treated with LED light device for 10 minutes, 4 times over the course of 2 months
  Arms: High intensity LED light treatment
Device: Sham LED light device — Participants have the light treatment moved off their wound after masking
  Arms: Sham high intensity LED light treatment

SUMMARY:
Diabetic and venous ulcers affect many people, and severe cases can end up in amputation and even death because of infection. In 2011, the total cost for care of diabetic foot ulcers alone, to the Canadian health care system, was $547 million. Standard clinical care for these types of wounds has improved but there is still a great need for new wound care treatments to help speed up wound healing and reduce pain. One such treatment is high intensity LED light therapy. There is a long history of light therapy showing faster wound healing, reduced pain and reduced swelling. The research we propose here is to study a new high intensity LED light made by Kerber Applied Research Inc., to see if it reduces pain and speeds up healing lower leg ulcers. This research is a partnership between Kerber Applied Research Inc and the Lethbridge Lower Limb Wound Clinic, an Alberta Health Services program in Lethbridge, Alberta.

DETAILED DESCRIPTION:
Purpose: To test the safety of a new LED light therapy device on patients with chronic diabetic or venous lower extremity ulcers, and to determine whether the light device decreases pain and accelerates wound healing.

Hypothesis: Patients with chronic diabetic or venous foot/leg ulcers treated with standard care plus 10 minutes of high intensity LED light therapy will experience less overall pain associated with their ulcer and the ulcer will heal faster than standard care alone.

Justification: Diabetic and venous foot ulcers are debilitating, costly, extremely painful and interfere significantly with quality of life. Standard care for chronic wounds has improved but there is great need of new treatments to complement wound care, reduce pain, and accelerate wound healing. High intensity LED light therapy is a re-emerging treatment option that is known to decrease inflammation, decrease pain, and increase tissue regeneration.

Objectives: The primary objective is to assess the safety of a high intensity LED light device (KPTL-10) in the treatment of chronic foot and leg ulcers. The secondary objectives are to assess the ability of the KPTL-10 device to reduce pain and accelerate wound healing.

Research Method/Procedures: Participants with chronic foot and leg ulcers less than 8 cm in diameter (longest direction) will randomized into one of 2 groups for this study: 1) to receive a free 10 minute light treatment with the KPTL10 device in addition to standard care, or 2) strictly be a part of the standard care control group (no light treatment). For treatment, the light device is placed at a fixed distance (1 cm) above the wound. All participants will have wound measurements taken with digital software throughout the course of the study to track wound healing. Patients will also record their pain levels by filling out a VAS pain scale throughout the study.

Plan for Data Analysis: For each study participant, detailed Case Report Forms will be completed by study researchers and the principal investigator Dr. Eric Bly at every study appointment. The target numbers for this study data set are 40 treated participants, and 20 control (untreated) participants. These case report forms contain data sections to capture wound sizes, patient experiences post treatment, and pain scores (VAS scale). All data will be stored digitally on a single study computer and manually as printed hardcopies for study records and complete data analysis by Dr. Eric Bly and Illumacell's clinical team.

ELIGIBILITY:
Inclusion Criteria:

* diabetic and venous lower limb ulcers less than or equal to 5cm in diameter
* healable wounds
* non-cancerous wounds

Exclusion Criteria:

* pregnant or breast feeding women
* participants taking photosensitive drugs for concomitant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Change in wound healing time | 4 months
  To determine whether high intensity LED therapy promotes changes in healing time of chronic foot ulcers. Participants will have the area (cm2) of their wounds calculated using Imitomeasure digital imaging software. Wound size will be tracked over the course of 4 light treatments.
Altered pain experience associated with chronic wounds | 4 months
  To determine whether high intensity LED therapy leads to altered pain experienced during standard care of chronic foot ulcers. Participants pain will be assessed by completing a pain questionnaire including the VAS pain scale measurement, over the course of 4 light treatments. Participants will complete the VAS pain scale measurement before and after each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Hummel, PhD, Study Director — Illumacell Inc.
Locations (1):
- Alberta Health Services - Lower Limb Wound Care, Lethbridge, Alberta, Canada

REFERENCES:
- See also: Website contains Abstract and Data Summary for "ILLUMACELL AND AHS PROFESSIONAL SUMMARY OF WOUND CARE ALBERTA (WCAB) STUDY" — http://www.illumacell.com